CLINICAL TRIAL: NCT03525444
Title: A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-445 Combination Therapy in Subjects With Cystic Fibrosis Who Are Heterozygous for the F508del Mutation and a Minimal Function Mutation (F/MF)
Brief Title: A Phase 3 Study of VX-445 Combination Therapy in Subjects With Cystic Fibrosis Heterozygous for the F508del Mutation and a Minimal Function Mutation (F/MF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX17-445-102; 2018-000183-28 (EudraCT Number)
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants who received placebo matched to VX-445/TEZ/IVA for 24 weeks in the TC treatment period.
  Interventions: Drug: Placebo
- VX-445/TEZ/IVA TC (Experimental): Participants who received VX-445 200 mg/TEZ 100 mg/IVA150 mg as fixed-dose combination (FDC) tablets in the morning and IVA 150 mg as mono tablet in the evening for 24 weeks in the TC treatment period.
  Interventions: Drug: VX-445/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: VX-445/TEZ/IVA — Participants received VX-445/TEZ/IVA orally once daily in the morning.
  Other Names: VX-445/VX-661/VX-770; VX-445/tezacaftor/ivacaftor
  Arms: VX-445/TEZ/IVA TC
Drug: IVA — Participants received IVA orally once daily in the evening
  Other Names: VX-770; ivacaftor
  Arms: VX-445/TEZ/IVA TC
Drug: Placebo — Participants received placebo matched VX-445/TEZ/IVA orally once daily in the morning and placebo matched to IVA orally once daily in the evening.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of VX-445 in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in subjects with cystic fibrosis (CF) who are heterozygous for F508del and a minimal function mutation (F/MF subjects).

ELIGIBILITY:
Key Inclusion Criteria:

* Heterozygous for the F508del mutation (F/MF)
* Forced expiratory volume in 1 second (FEV1) value ≥40% and ≤90% of predicted mean for age, sex, and height

Key Exclusion Criteria:

* Clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Solid organ or hematological transplantation

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (115):
- United States (53):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Miller Children's Hospital/ Long Beach Memorial, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital/ Children's Hospital of Central California, Madera, California
  - Kaiser Permanente, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Gateway Medical Center, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - University of Florida, Shands Hospital, Gainesville, Florida
  - Joe DiMaggio Cystic Fibrosis & Pulmonary Center/ Joe DiMaggio Children's Hospital/ Memorial Regional Hospital, Hollywood, Florida
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Tampa General Hospital Cardiac and Lung Transplant Clinic, Tampa, Florida
  - Children's Speciality Services at North Druid Hills, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Saint Francis Medical Center/ Children's Hospital of Illinois/OSF, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane Medical Center, New Orleans, Louisiana
  - Maine Medical Partners, Portland, Maine
  - Massachusetts General Hospital Cystic Fibrosis Center, Boston, Massachusetts
  - Harper University Hospital, Detroit, Michigan
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Billings Clinic, Billings, Montana
  - Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - University of New Mexico Clinical & Translational Science Center, Albuquerque, New Mexico
  - Mount Sinai Beth Israel, New York, New York
  - New York Medical College, Valhalla, New York
  - UNC Marsico Clinical Research Center, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - UC Health Holmes, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center/ Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/ Toledo Children's Hospital/ Pediatric Pulmonary & Cystic Fibrosis Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Austin Children's Chest Associates, Austin, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - Vermont Lung Center, Colchester, Vermont
  - University of Virginia Primary Care Center, Charlottesville, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Hospital of Richmond at VCU, Children's Pavilion, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
  - CTSI Adult Translational Research Unit/Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Australia (5):
  - Women & Children's Hospital, North Adelaide
  - The Royal Children's Hospital, Parkville
  - Mater Adult Hospital, South Brisbane
  - The Children's Hospital at Westmead, Westmead
  - Westmead Hospital, Westmead
- Austria (4):
  - University of Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Medizinische Universitat Wien, Vienna
- Belgium (5):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gathuisberg, Leuven
- Canada (8):
  - British Columbia's Children's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal, Quebec
  - University of Calgary Medical Clinic of the Foothills Medical Centre, Calgary
  - Centre Hospitalier De L'Universite Laval, Qubec
  - Saint John Regional Hospital, Saint John
  - The Hospital for Sick Children, Toronto
  - Vancouver Island Health Authority, Victoria
- Czechia (2):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni nemocnice v Motole, Prague
- France (7):
  - Centre Hospitalier Lyon Sud, Benite Cedex
  - Groupe Hospitaler Pellegrin, CHU De Bordeaux, Bordeaux
  - CHU Marseille - Hopital Nord, Marseille
  - CHU de Nice - Hopital Pasteur, Nice
  - Hopital Cochin, Paris
  - CHU de Rouen - Hopital Charles Nicolle, Rouen Cedex, Seine Maritime
  - Hopital Foch (Suresnes), Hopital Foch, Adultes, Suresnes
- Germany (8):
  - Friedrich-Alexander University of Erlangen-Nuremberg, University Children's Hospital, Erlangen
  - Justus-Leibig-Universitat Zentrum fur Kinderheilkunde und Jugendmedizin, Giessen
  - Hannover Medical School, Hanover
  - Heidelberg Cystic Fibrosis Center, Heidelberg
  - Johannes Gutenberg-Universitaet, Mainz
  - Dr. von Haunersches Kinderspital, München
  - Universitaetsklinikum Tuebingen Klinik fuer Kinder- und Jugendmedizin, Tübingen
  - University Hospital Wuerzburg, Würzburg
- General Hospital of Attika "Sismanoglio"(Adult CF center, NHS), Marousi, Greece
- Italy (7):
  - Azienda Ospedaliero Universitaria Ospedale Riuniti, Ancona
  - Azienda Ospedaliero Universitaria Ospedale Pediatrico Meyer, Florence
  - IRCCS Istituto Giannina Gaslini-Ospedale Pediatrico, Genova
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Centro Regionale Fibrosi Cistica, A.O. Ospedale San Carlo, Potenza
  - Azienda Ospedaliera di Verona-Ospedale Civile Maggiore, Verona
- Netherlands (5):
  - Academic Medical Center, Amsterdam
  - University Medical Center, Utrecht, Department of Pulmonology and Tuberculosis, Heidelberglaan
  - UMC St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis van den Haag, The Hague
- Karolinska Univeritetssjukhuset, Huddinge, Stockholm, Sweden
- United Kingdom (9):
  - The Royal Belfast Hospital for Sick Children, Belfast
  - Heart of England NHS Foundation Trust, Birmingham Heartlands Hospital, Brimingham
  - Royal Hospital for Sick Children, Edinburgh
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter NHS Foundation Trust, Royal Devon and Exeter Hospital, Exeter
  - Leeds General Infirmary, Leeds
  - King's College Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Middleton PG, Mall MA, Drevinek P, Lands LC, McKone EF, Polineni D, Ramsey BW, Taylor-Cousar JL, Tullis E, Vermeulen F, Marigowda G, McKee CM, Moskowitz SM, Nair N, Savage J, Simard C, Tian S, Waltz D, Xuan F, Rowe SM, Jain R; VX17-445-102 Study Group. Elexacaftor-Tezacaftor-Ivacaftor for Cystic Fibrosis with a Single Phe508del Allele. N Engl J Med. 2019 Nov 7;381(19):1809-1819. doi: 10.1056/NEJMoa1908639. Epub 2019 Oct 31. PMID 31697873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 405 participants were enrolled in the study, of which 2 participants were enrolled but were not dosed in the triple combination (TC) treatment period. Results are presented for 403 participants dosed in the TC treatment period.
Pre-assignment Details: This study was conducted in participants with cystic fibrosis (CF) aged 12 years or older.
Groups:
- Placebo: Participants who received placebo matched to VX-445/TEZ/IVA in the morning and placebo matched to IVA in the evening for 24 weeks in the TC treatment period.
Period: Overall Study
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Started | 203 | 200
Safety Set (Based on actual treatment received.) | 201 | 202
Completed | 203 | 197
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal of consent (not due to AE) | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who carried the intended CF transmembrane conductance regulator gene (CFTR) allele mutation and received at least 1 dose of study drug in the TC Treatment Period.
Groups:
- VX-445/TEZ/IVA TC: Participants who received VX-445 200 mg/TEZ 100 mg/IVA150 mg as FDC tablets in the morning and IVA 150 mg as mono tablet in the evening for 24 weeks in the TC treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | VX-445/TEZ/IVA TC | Total
Number analyzed (Participants) | 203 | 200 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (11.3) | 25.6 (9.7) | 26.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 96 | 194
  Male | 105 | 104 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 4 | 16
  Not Hispanic or Latino | 175 | 187 | 362
  Unknown or Not Reported | 16 | 9 | 25
Race [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Black or African American | 1 | 3 | 4
  Not Collected per Local Regulations | 16 | 9 | 25
  Australian Aboriginal | 0 | 1 | 1
  Not Otherwise Specified | 1 | 0 | 1
  Other- Unknown Mixed Heritage | 0 | 1 | 1
  White | 182 | 185 | 367
  White, Asian | 1 | 0 | 1
  White, Black or African American | 1 | 1 | 2
Forced Expiratory Volume in 1 Second (ppFEV1) [Mean (Standard Deviation); unit: percentage points] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
  percentage points | 61.3 (15.5) | 61.6 (15.0) | 61.4 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline at Week 4
Population: Analysis population included all participants in the Full Analysis Set (all randomized participants who carried the intended CFTR allele mutation and received at least 1 dose of study drug) who completed the Week 4 Visit or were randomized at least 28 days before the data cutoff date.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 203 | 200
percentage points | -0.2 (0.6) | 13.6 (0.6)
Statistical Analysis 1: Comparison: Placebo vs VX-445/TEZ/IVA TC; The data presented for Primary endpoint was based on interim analysis at Week 4; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; Least Squares (LS) Mean Difference = 13.8, 95% CI 2-sided [12.1 to 15.4]

2. Secondary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 203 | 200
percentage points | -0.4 (0.5) | 13.9 (0.6)
Statistical Analysis 1: Comparison: Placebo vs VX-445/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = 14.3, 95% CI 2-sided [12.7 to 15.8]

3. Secondary Outcome: Number of Pulmonary Exacerbations (PEx)
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms.
Time Frame: From Baseline through Week 24
Population: FAS.
Measure: Number; unit: pulmonary exacerbation events
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 203 | 200
pulmonary exacerbation events | 113 | 41
Statistical Analysis 1: Comparison: Placebo vs VX-445/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Negative binomial regression model; Rate ratio = 0.37, 95% CI 2-sided [0.25 to 0.55]

4. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline through Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 203 | 200
millimole per liter (mmol/L) | -0.4 (0.9) | -42.2 (0.9)
Statistical Analysis 1: Comparison: Placebo vs VX-445/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = -41.8, 95% CI 2-sided [-44.4 to -39.3]

5. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline through Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 203 | 200
units on a scale | -2.7 (1.0) | 17.5 (1.0)
Statistical Analysis 1: Comparison: Placebo vs VX-445/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = 20.2, 95% CI 2-sided [17.5 to 23.0]

6. Secondary Outcome: Absolute Change in Body Mass Index (BMI)
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2).
Time Frame: From Baseline at Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: kilogram per meter square (kg/m^2)
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 203 | 200
kilogram per meter square (kg/m^2) | 0.09 (0.07) | 1.13 (0.07)
Statistical Analysis 1: Comparison: Placebo vs VX-445/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = 1.04, 95% CI 2-sided [0.85 to 1.23]

7. Secondary Outcome: Absolute Change in Sweat Chloride
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline at Week 4
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 203 | 200
mmol/L | 0.1 (1.0) | -41.2 (1.0)
Statistical Analysis 1: Comparison: Placebo vs VX-445/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = -41.2, 95% CI 2-sided [-44.0 to -38.5]

8. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire Revised (CFQ-R) Respiratory Domain Score
Description: as for outcome 5
Time Frame: From Baseline at Week 4
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 203 | 200
units on a scale | -1.9 (1.1) | 18.1 (1.1)
Statistical Analysis 1: Comparison: Placebo vs VX-445/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = 20.1, 95% CI 2-sided [16.9 to 23.2]

9. Secondary Outcome: Time-to-first Pulmonary Exacerbation (PEx)
Description: as for outcome 3
Time Frame: From Baseline through Week 24
Population: FAS.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 203 | 200
days | NA [NA to NA] — Median and 95% confidence interval could not be estimated because less than 50% of participants had events. | NA [NA to NA] — Median and 95% confidence interval could not be estimated because less than 50% of participants had events.

10. Secondary Outcome: Absolute Change in BMI Z-score for Participants <=20 Years of Age at Baseline
Description: BMI was defined as weight in kg divided by height in m^2. Z-score is a statistical measure to describe whether a mean was above or below the standard. BMI, adjusted for age and sex, was analyzed as BMI-for-age z-score. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of higher BMI.
Time Frame: From Baseline at Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were <=20 years of age at Baseline.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 74 | 71
z-score | 0.04 (0.05) | 0.34 (0.05)
Statistical Analysis 1: Comparison: Placebo vs VX-445/TEZ/IVA TC; Test type: Superiority; LS Mean Difference = 0.30, 95% CI 2-sided [0.17 to 0.43]

11. Secondary Outcome: Absolute Change in Body Weight
Time Frame: From Baseline at Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 203 | 200
kg | 0.5 (0.2) | 3.4 (0.2)
Statistical Analysis 1: Comparison: Placebo vs VX-445/TEZ/IVA TC; Test type: Superiority; LS Mean Difference = 2.9, 95% CI 2-sided [2.3 to 3.4]

12. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug or to the completion of study participation date, whichever occurs first (up to 28 weeks)
Population: Adverse events are presented as per Safety Set. Group assignments for participants in the Safety Set were based on actual treatment received, such that 2 participants assigned to Placebo group who inadvertently received one or more doses of VX-445/TEZ/IVA TC regimen were included in VX-445/TEZ/IVA TC group for the purpose of safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 201 | 202
Participants
  Participants with TEAEs | 193 | 188
  Participants with Serious TEAEs | 42 | 28

13. Secondary Outcome: Observed Pre-dose Concentration (Ctrough) of VX-445, TEZ, M1-TEZ, and IVA
Time Frame: Pre-dose on Week 4, 8, 12, and 16
Population: Pharmacokinetic (PK) set included all randomized participants who carried the intended CFTR allele mutation and received at least 1 dose of study drug in the TC Treatment Period. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 200
microgram per milliliter (mcg/mL)
  VX-445 (Week 4): number analyzed (Participants) | 198
  VX-445 (Week 4) | 5.02 (2.68)
  VX-445 (Week 8): number analyzed (Participants) | 192
  VX-445 (Week 8) | 4.90 (2.75)
  VX-445 (Week 12): number analyzed (Participants) | 195
  VX-445 (Week 12) | 4.99 (3.11)
  VX-445 (Week 16): number analyzed (Participants) | 196
  VX-445 (Week 16) | 4.75 (2.58)
  TEZ (Week 4): number analyzed (Participants) | 198
  TEZ (Week 4) | 2.16 (1.05)
  TEZ (Week 8): number analyzed (Participants) | 193
  TEZ (Week 8) | 2.14 (1.14)
  TEZ (Week 12): number analyzed (Participants) | 196
  TEZ (Week 12) | 2.22 (1.48)
  TEZ (Week 16): number analyzed (Participants) | 196
  TEZ (Week 16) | 2.32 (1.46)
  M1-TEZ (Week 4): number analyzed (Participants) | 198
  M1-TEZ (Week 4) | 5.18 (2.01)
  M1-TEZ (Week 8): number analyzed (Participants) | 193
  M1-TEZ (Week 8) | 5.09 (1.95)
  M1-TEZ (Week 12): number analyzed (Participants) | 196
  M1-TEZ (Week 12) | 5.06 (1.92)
  M1-TEZ (Week 16): number analyzed (Participants) | 196
  M1-TEZ (Week 16) | 5.29 (1.95)
  IVA (Week 4): number analyzed (Participants) | 197
  IVA (Week 4) | 0.748 (0.471)
  IVA (Week 8): number analyzed (Participants) | 193
  IVA (Week 8) | 0.738 (0.484)
  IVA (Week 12): number analyzed (Participants) | 196
  IVA (Week 12) | 0.758 (0.572)
  IVA (Week 16): number analyzed (Participants) | 196
  IVA (Week 16) | 0.778 (0.516)

ADVERSE EVENTS:
Time Frame: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug or to the completion of study participation date, whichever occurs first (up to 28 weeks)
Description: Adverse events are presented as per Safety Set. Group assignments for participants in the Safety Set were based on actual treatment received, such that 2 participants assigned to Placebo group who inadvertently received one or more doses of VX-445/TEZ/IVA TC regimen were included in VX-445/TEZ/IVA TC group for the purpose of safety analysis.
Arm/Group | Placebo | VX-445/TEZ/IVA TC
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/202
Serious Adverse Events (participants affected / at risk) | 42/201 | 28/202
Other Adverse Events (participants affected / at risk) | 180/201 | 168/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=201) | VX-445/TEZ/IVA TC (N=202)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 33 | 11
Influenza (Infections and infestations) | 0 | 3
Atypical mycobacterial lower respiratory tract infection (Infections and infestations) | 1 | 0
Coccidioidomycosis (Infections and infestations) | 1 | 0
Genital herpes simplex (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Viral sinusitis (Infections and infestations) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Gallbladder enlargement (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Axonal neuropathy (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 1
Neuroglycopenia (Nervous system disorders) | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1
Medical device site inflammation (General disorders) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=201) | VX-445/TEZ/IVA TC (N=202)
Cough (Respiratory, thoracic and mediastinal disorders) | 77 | 34
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 39 | 40
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 | 20
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 27 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 | 19
Productive cough (Respiratory, thoracic and mediastinal disorders) | 16 | 12
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 5
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 83 | 41
Nasopharyngitis (Infections and infestations) | 26 | 22
Upper respiratory tract infection (Infections and infestations) | 22 | 24
Rhinitis (Infections and infestations) | 11 | 15
Sinusitis (Infections and infestations) | 8 | 11
Influenza (Infections and infestations) | 3 | 12
Diarrhoea (Gastrointestinal disorders) | 14 | 26
Abdominal pain (Gastrointestinal disorders) | 12 | 20
Nausea (Gastrointestinal disorders) | 14 | 16
Vomiting (Gastrointestinal disorders) | 10 | 12
Constipation (Gastrointestinal disorders) | 12 | 6
Alanine aminotransferase increased (Investigations) | 7 | 20
Blood creatine phosphokinase increased (Investigations) | 9 | 19
Aspartate aminotransferase increased (Investigations) | 4 | 19
Bacterial test positive (Investigations) | 10 | 5
Blood bilirubin increased (Investigations) | 2 | 10
Headache (Nervous system disorders) | 30 | 35
Pyrexia (General disorders) | 19 | 17
Fatigue (General disorders) | 20 | 9
Rash (Skin and subcutaneous tissue disorders) | 9 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT03525444/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT03525444/SAP_001.pdf